CLINICAL TRIAL: NCT00217880
Title: Prognostic Significance of Biological Markers in Patients With ALI/ARDS
Brief Title: Significance of Biological Markers in Patients With Acute Lung Injury/Acute Respiratory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Theodore J. Standiford, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 292; P50HL074024 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2009-07

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bronchoscopy — A bronchoscopy test will occur to view the participant's airways.

SUMMARY:
The purpose of this study is to identify biological markers of disease in patients with acute lung injury (ALI) that are predictive of either disease susceptibility or prognosis, or that identify novel targets of therapeutic intervention.

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory failure due to ALI and acute respiratory distress syndrome (ARDS) remains a major health problem despite significant progress in intensive care unit (ICU) care and ventilator management. It is also characterized by an unacceptably high mortality rate despite enormous expenditure of health care resources. Survivors of respiratory failure face long-term consequences concerning their quality of life. New therapies are needed to improve early survival and to decrease long-term sequelae of this syndrome. The purpose of this study is to identify biological markers of disease in patients with ALI that are predictive of either disease susceptibility or prognosis, or that identify novel targets of therapeutic intervention.

DESIGN NARRATIVE:

As soon as possible after case identification, informed consent will be obtained from the patient or next of kin. Physiologic measurements and specimen collection will begin at the time of entry into the study. The inclusion criteria for this study allow entry of patients who have fulfilled criteria for ALI/ARDS for up to 48 hours. Bronchoalveolar lavage (BAL) fluid and blood will be collected at various times after the onset of ALI/ARDS in order to measure levels of a predetermined set of biological markers. In addition, DNA will be collected from patients and analysed for the presence of specific genetic polymorphisms that might alter either disease susceptibility or clinical expression of disease. The levels of these markers or the presence of specific genetic polymorphisms will be correlated with measure of pulmonary inflammation and extent of lung injury, as defined by: 1) PaO2/FiO2 ratios; 2) lung compliance; 3) plateau pressures; and 4) calculation of the Murray Lung Injury Score (obtained at entry and Days 1, 2, 3, 5, 7,10, 14, and 21). Secondary outcome measures to be directly correlated with biomarker expression will include indicators of maladaptive responses to ALI (including the development of multiple organ dysfunction syndrome [MODS]), fibroproliferation, and nosocomial pneumonia (events which greatly impact the clinical course of patients with ALI/ARDS). Thus, the secondary outcome measures include: 1) the development of organ failure (using the Sequential Organ Failure Assessment [SOFA] score); 2) time on ventilator; 3) ventilator-free days; 4) ICU and hospital length of stay; 5) hospital mortality; 6) development of pneumonia; 7) development of lung fibrosis (as determined by high-resolution computed tomography [HRCT] and pulmonary function testing); and 8) health related and lung-specific quality of life (as assessed with the Medical Outcome Studies 36-Item Short form Health Survey Standard Form [SF-36] and St. George's Respiratory Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

Acute onset of illness with:

* PaO2/FiO2 ratio of less than 300 (ALI) or PaO2/FiO2 ratio of less than 200 (ARDS)
* Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph (infiltrates may be patchy, diffuse, homogeneous, or asymmetric)
* Positive pressure ventilation via an endotracheal tube
* No clinical evidence of left atrial hypertension (if measured, pulmonary arterial wedge pressure less than or equal to 18 mm Hg)
* First three criteria must occur together within a 24-hour interval

Exclusion Criteria:

* Greater than 48 hours elapsed following institution of mechanical ventilation
* Pregnancy
* Chronic respiratory failure as defined by any of the following:

  1. FEV1 less than 20 ml/kg of PBW; FEV1/FVC less than 50%
  2. Chronic hypercapnia or hypoxemia
  3. Hospitalization within past 6 months for acute respiratory failure
  4. Chronic home use of oxygen or mechanical ventilation
* Left ventricular failure as defined by New York Heart Association (NYHA) class IV status
* History of hematological malignancy or bone marrow transplantation
* Entry in other intervention clinical trials
* Decision of the patient or attending physician to forego aggressive care
* Expected survival of less than 6 months (based solely on pre-existing medical problems [e.g., poorly controlled neoplasm or other end-stage disease])
* AIDS (known history of HIV infection)
* Prednisone (or equivalent) therapy of 20 mg/day or more for a period of at least 2 months with treatment continuing within 3 weeks prior to screening
* Cytotoxic therapy within 3 weeks of screening
* Morbid obesity defined as greater than 1 kg/c body weight
* At risk for increased intracranial pressure that may result from permissive hypercapnia
* Permissive hypercapnia that is contraindicated
* Neuromuscular disease that would potentially impact ability to wean from mechanical ventilation
* Receiving extracorporeal membrane oxygenation when meeting screening criteria

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-07; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratios | Measured at Year 4
Lung compliance | Measured at Year 4
Plateau pressures | Measured at Year 4
Calculation of the Murray Lung Injury Score (obtained at entry and Days 1, 2, 3, 5, 7,10, 14, and 21; analyzed at Year 4) | Measured at Year 4

SECONDARY OUTCOMES:
Development of organ failure | Measured at Year 4
Time on ventilator | Measured at Year 4
Ventilator-free days | Measured at Year 4
ICU and hospital length of stay | Measured at Year 4
Hospital mortality | Measured at Year 4
Development of pneumonia | Measured at Year 4
Development of lung fibrosis | Measured at Year 4
Health-related and lung-specific quality of life | Measured at Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Theodore J. Standiford, MD, Study Chair — University of Michigan
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan